CLINICAL TRIAL: NCT04963231
Title: A 2-Stage (Open-Label Followed by Randomized Double-Blind, Placebo-Controlled Stage), Phase 2 Trial of Setmelanotide in Patients With Specific Gene Variants in the Melanocortin-4 Receptor Pathway
Brief Title: DAYBREAK: A Study of Setmelanotide in Participants With Specific Gene Variants in the Melanocortin-4 Receptor (MC4R) Pathway
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM-493-034
Record Dates: First submitted 2021-06-28; First posted 2021-07-15 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Genetic Obesity
Keywords: Melanocortin-4 Receptor; Genetic Obesity; Leptin
MeSH Terms: interventions — setmelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Stage 1 of the trial is open-label. Participants who were eligible to enter Stage 2 of the trial were randomized in a blinded manner at the Stage 2 Entry Visit in a 2:1 ratio to receive either setmelanotide or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Stage 1: Setmelanotide (Open-Label) (Experimental): Participants received once daily SC injection of setmelanotide from Day 1 to Week 16 in an open-label treatment stage (Stage 1). Participants ≥12 years of age started on setmelanotide 2.0 milligrams (mg) once daily for approximately 2 weeks, then increased to 3.0 mg once daily. Participants <12 years of age started on setmelanotide 1.0 mg once daily for approximately 1 week, then increased to 2.0 mg once daily for approximately 1 week, then increased to 3.0 mg once daily.
  Interventions: Drug: Setmelanotide
- Stage 2: Setmelanotide (Double-Blind) (Experimental): Participants from Stage 1 who were eligible for Stage 2 received once daily SC injection of setmelanotide 3.0 mg from Week 16 to Week 40 in a double-blind treatment Stage (Stage 2).
  Interventions: Drug: Setmelanotide
- Stage 2: Placebo (Double-Blind) (Placebo Comparator): Participants from Stage 1 who were eligible for Stage 2 received once daily SC injection of matching placebo 3.0 mg from Week 16 to Week 40 in a double-blind treatment Stage (Stage 2).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Setmelanotide — SC injection
  Arms: Stage 1: Setmelanotide (Open-Label); Stage 2: Setmelanotide (Double-Blind)
Drug: Placebo — SC injection
  Arms: Stage 2: Placebo (Double-Blind)

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of once daily subcutaneous (SC) administration of setmelanotide in participants with obesity and specific gene variants in the MC4R pathway.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have had a pre-identified genetic variant in an established MC4R pathway gene that contributes to obesity
* Age 6 to 65 years, inclusive
* Obesity, defined as Body Mass Index (BMI) ≥40 kilograms per square meter (kg/m^2) for participants ≥18 years of age or BMI ≥97th percentile for age and gender for participants 6 to <18 years of age
* Study participant and/or parent or guardian were able to understand all study procedures and provide consent/assent
* Use of highly effective contraception
* Symptoms or behaviors of hyperphagia

Key Exclusion Criteria:

* Participants with the following genetic variants: biallelic Bardet-Biedl Syndrome (BBS); biallelic Alström Syndrome 1 (ALMS1); homozygous, heterozygous, or compound heterozygous variants in MC4R, Pro-opiomelanocortin (POMC), Proprotein convertase subtilisin/kexin type 1 (PCSK1), Leptin receptor (LEPR), nuclear receptor coactivator 1 (NCOA1; steroid receptor coactivator-1 [SRC1]) or SRC homology 2 B adapter protein 1 (SH2B1) genes as well as 16p11.2 chromosomal deletions that included the SH2B1 gene
* Recent intensive diet and/or exercise regimen with or without the use of weight loss agents including herbal medications that had resulted in weight loss >2% within previous 3 months
* Bariatric surgery within the previous 6 months
* Documented diagnosis of current unstable major psychiatric disorder or a documented worsening of psychiatric condition that required changes in treatment within 2 years
* Any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) or Patient Health Questionnaire 9 (PHQ 9) score of ≥15 during Screening, any suicide attempt in participant's lifetime years, or any suicidal behavior in the last month.
* Current, clinically significant pulmonary, cardiac, or oncologic disease considered severe enough to interfere with the study
* Has significant features of (or meets the diagnostic criteria for) a genetic syndrome that is associated with obesity
* Glycated hemoglobin (HbA1C) >10.0% at Screening
* History of significant liver disease
* Glomerular filtration rate (GFR) <30 milliliter per minute (mL/min) at Screening
* History or close family history of melanoma or participant history of oculocutaneous albinism
* Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions
* Participation in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing
* Participants previously enrolled in a clinical study involving setmelanotide or any previous exposure to setmelanotide
* Significant hypersensitivity to any excipient in the study drug
* Females who were breastfeeding or nursing

Other protocol defined Inclusion/Exclusion criteria applied.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (36):
- United States (21):
  - HonorHealth Bariatric Center, Scottsdale, Arizona
  - InQuest Medical Reseacrh, Suwanee, Georgia
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Metro Detroit Endocrinology Center, Dearborn, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - Ten's Medical Center - Pediatric Endocrinology Clinic, Staten Island, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Geisinger Clinic, Danville, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Tech, Amarillo, Texas
  - Endocrine Associates of Dallas and Plano, Dallas, Texas
  - Hector Granados PA, El Paso, Texas
  - Texas Children's Hospital, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Rio Grande Valley Endocrine Center, McAllen, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Javara Research, The Woodlands, Texas
- University of Alberta, Edmonton, Alberta, Canada
- Germany (3):
  - Charite - Universitatsmedizin Berlin, Berlin
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Ulm, Ulm
- University of Patras School of Medicine, Pátrai, Greece
- Chaim Sheba MC, Safra Children's Hospital, Ramat Gan, Israel
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Spain (4):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Fundación Jimenez Díaz, Madrid
  - Hospital General de Valencia, Valencia
- United Kingdom (4):
  - Bristol Royal Hospital for Children, Bristol
  - University of Cambridge, Cambridge
  - London Medical - The London Diabetes Centre, London
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trapp CM, Censani M. Setmelanotide: a promising advancement for pediatric patients with rare forms of genetic obesity. Curr Opin Endocrinol Diabetes Obes. 2023 Apr 1;30(2):136-140. doi: 10.1097/MED.0000000000000798. Epub 2023 Feb 1. PMID 36722447
- [Derived] Cuda S, Censani M. Progress in pediatric obesity: new and advanced therapies. Curr Opin Pediatr. 2022 Aug 1;34(4):407-413. doi: 10.1097/MOP.0000000000001150. Epub 2022 Jul 5. PMID 35797460

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 218 participants were screened and 164 participants received at least one dose of trial medication in Stage 1.
Groups:
- Stage 1: Setmelanotide (Open-Label): Participants received once daily subcutaneous (SC) injection of setmelanotide from Day 1 to Week 16 in an open-label treatment stage (Stage 1). Participants ≥12 years of age started on setmelanotide 2.0 milligrams (mg) once daily for approximately 2 weeks, then increased to 3.0 mg once daily. Participants <12 years of age started on setmelanotide 1.0 mg once daily for approximately 1 week, then increased to 2.0 mg once daily for approximately 1 week, then increased to 3.0 mg once daily.
Period: Stage 1 (Open-Label, Duration: 16 Weeks)
Arm/Group | Stage 1: Setmelanotide (Open-Label) | Stage 2: Setmelanotide (Double-Blind) | Stage 2: Placebo (Double-Blind)
Started | 164 | 0 | 0
Completed | 100 | 0 | 0
Not Completed | 64 | 0 | 0
Not completed — Adverse Event | 43 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Period: Stage 2 (Double-Blind, Duration:24 Week)
Arm/Group | Stage 1: Setmelanotide (Open-Label) | Stage 2: Setmelanotide (Double-Blind) | Stage 2: Placebo (Double-Blind)
Started (Participants who completed Stage 1 were assessed for eligibility in Stage 2. At the Stage 2 Entry Visit, all eligible participants were randomized 2:1 to either continue daily setmelanotide or receive matching placebo.) | 0 | 32 | 17
Safety Analysis Set Enrolled in Stage 2 (All participants who were enrolled in Stage 2 and received at least one dose of trial medication in Stage 2. Three participants in the placebo group were rescued with setmelanotide open-label during Stage 2. They were classified to setmelanotide group.) | 0 | 35 | 14
Completed | 0 | 29 | 10
Not Completed | 0 | 3 | 7
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Other than specified | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least one dose of trial medication.
Groups:
- All Participants: Stage 1: All participants received once daily SC injection of setmelanotide for 16 weeks in an open-label treatment Stage. Participants ≥12 years of age started on setmelanotide 2.0 mg once daily for approximately 2 weeks, then increased to 3.0 mg once daily. Participants <12 years of age started on setmelanotide 1.0 mg once daily for approximately 1 week, then increased to 2.0 mg once daily for approximately 1 week, then increased to 3.0 mg once daily.
  Stage 2: Participants from Stage 1 who were eligible for Stage 2 received once daily SC injection of setmelanotide 3.0 mg or matching placebo from Week 16 to Week 40 in a double-blind treatment Stage.
Arm/Group | All Participants
Number analyzed (Participants) | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (16.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 124
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 128
  More than one race | 0
  Unknown or Not Reported | 16

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Number of Participants by Genotype Who Demonstrated a Significant Clinically Meaningful Response to Setmelanotide at the End of Stage 1
Description: BMI was calculated using participant's weight and height assessments, using the following formula: BMI = Kilogram (kg)/ square meter (m^2).
  A significant clinically meaningful response was defined as achieving a ≥5% reduction in BMI from Baseline.
  Data are provided for overall and according to participants with specified primary gene. Baseline was defined as the last available measurement taken prior to the start of treatment Stage 1 administration.
Time Frame: Baseline to Week 16
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Stage 1: Setmelanotide (Open-Label): Participants received once daily SC injection of setmelanotide from Day 1 to Week 16 in an open-label treatment stage (Stage 1). Participants ≥12 years of age started on setmelanotide 2.0 mg once daily for approximately 2 weeks, then increased to 3.0 mg once daily. Participants <12 years of age started on setmelanotide 1.0 mg once daily for approximately 1 week, then increased to 2.0 mg once daily for approximately 1 week, then increased to 3.0 mg once daily.
Arm/Group | Stage 1: Setmelanotide (Open-Label)
Number analyzed (Participants) | 164
Participants
  Overall | 49
  Gene: NRP1: number analyzed (Participants) | 2
  Gene: NRP1 | 0
  Gene: NRP2: number analyzed (Participants) | 3
  Gene: NRP2 | 0
  Gene: PLXNA1: number analyzed (Participants) | 8
  Gene: PLXNA1 | 2
  Gene: PLXNA2: number analyzed (Participants) | 9
  Gene: PLXNA2 | 3
  Gene: PLXNA3: number analyzed (Participants) | 3
  Gene: PLXNA3 | 2
  Gene: PLXNA4: number analyzed (Participants) | 20
  Gene: PLXNA4 | 5
  Gene: SEMA3A: number analyzed (Participants) | 3
  Gene: SEMA3A | 2
  Gene: SEMA3B: number analyzed (Participants) | 3
  Gene: SEMA3B | 1
  Gene: SEMA3C: number analyzed (Participants) | 1
  Gene: SEMA3C | 0
  Gene: SEMA3D: number analyzed (Participants) | 4
  Gene: SEMA3D | 0
  Gene: SEMA3E: number analyzed (Participants) | 6
  Gene: SEMA3E | 3
  Gene: SEMA3F: number analyzed (Participants) | 4
  Gene: SEMA3F | 2
  Gene: SEMA3G: number analyzed (Participants) | 24
  Gene: SEMA3G | 8
  Gene: PHIP: number analyzed (Participants) | 16
  Gene: PHIP | 9
  Gene: SIM1: number analyzed (Participants) | 20
  Gene: SIM1 | 5
  Gene: MAGEL2: number analyzed (Participants) | 10
  Gene: MAGEL2 | 3
  Gene: CREBBP: number analyzed (Participants) | 1
  Gene: CREBBP | 0
  Gene: DNMT3A: number analyzed (Participants) | 1
  Gene: DNMT3A | 0
  Gene: HTR2C: number analyzed (Participants) | 3
  Gene: HTR2C | 0
  Gene: KSR2: number analyzed (Participants) | 11
  Gene: KSR2 | 1
  Gene: MRAP2: number analyzed (Participants) | 1
  Gene: MRAP2 | 0
  Gene: RPGRIP1L: number analyzed (Participants) | 3
  Gene: RPGRIP1L | 1
  Gene: TBX3: number analyzed (Participants) | 5
  Gene: TBX3 | 2
  Gene: TRPC5: number analyzed (Participants) | 3
  Gene: TRPC5 | 0

2. Secondary Outcome: Mean Change in BMI From Baseline to the End of Stage 1 in All Participants, Per Genotype
Description: BMI was calculated using participant's weight and height assessments, using the following formula: BMI = kg/m^2.
  Data are provided for overall and according to participants with specified primary gene.
  Baseline was defined as the last available measurement taken prior to the start of treatment Stage 1 administration.
Time Frame: Baseline, Week 16
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Stage 1: Setmelanotide (Open-Label)
Number analyzed (Participants) | 164
Kg/m^2
  Overall: At Baseline | 45.338 (9.5526)
  Overall: Change at Week 16: number analyzed (Participants) | 112
  Overall: Change at Week 16 | -1.916 (1.7971)
  Gene: NRP1, At Baseline: number analyzed (Participants) | 2
  Gene: NRP1, At Baseline | 48.601 (2.7893)
  Gene: NRP1, Change at Week 16: number analyzed (Participants) | 2
  Gene: NRP1, Change at Week 16 | 0.229 (1.6024)
  Gene: NRP2, At Baseline: number analyzed (Participants) | 3
  Gene: NRP2, At Baseline | 46.568 (10.6754)
  Gene: NRP2, Change at Week 16: number analyzed (Participants) | 3
  Gene: NRP2, Change at Week 16 | -1.040 (0.8650)
  Gene: PLXNA1, At Baseline: number analyzed (Participants) | 8
  Gene: PLXNA1, At Baseline | 45.576 (5.5644)
  Gene: PLXNA1, Change at Week 16: number analyzed (Participants) | 5
  Gene: PLXNA1, Change at Week 16 | -1.884 (1.8912)
  Gene: PLXNA2, At Baseline: number analyzed (Participants) | 9
  Gene: PLXNA2, At Baseline | 48.577 (12.1795)
  Gene: PLXNA2, Change at Week 16: number analyzed (Participants) | 6
  Gene: PLXNA2, Change at Week 16 | -2.492 (2.0273)
  Gene: PLXNA3, At Baseline: number analyzed (Participants) | 3
  Gene: PLXNA3, At Baseline | 34.083 (6.4705)
  Gene: PLXNA3, Change at Week 16: number analyzed (Participants) | 2
  Gene: PLXNA3, Change at Week 16 | -3.333 (0.5166)
  Gene: PLXNA4, At Baseline: number analyzed (Participants) | 20
  Gene: PLXNA4, At Baseline | 46.634 (8.5714)
  Gene: PLXNA4, Change at Week 16: number analyzed (Participants) | 14
  Gene: PLXNA4, Change at Week 16 | -2.218 (2.9947)
  Gene: SEMA3A, At Baseline: number analyzed (Participants) | 3
  Gene: SEMA3A, At Baseline | 39.405 (7.8242)
  Gene: SEMA3A, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3A, Change at Week 16 | -2.328 (0.2612)
  Gene: SEMA3B, At Baseline: number analyzed (Participants) | 3
  Gene: SEMA3B, At Baseline | 42.890 (5.0100)
  Gene: SEMA3B, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3B, Change at Week 16 | -2.557
  Gene: SEMA3C, At Baseline: number analyzed (Participants) | 1
  Gene: SEMA3C, At Baseline | 47.543
  Gene: SEMA3C, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3C, Change at Week 16 | -2.334
  Gene: SEMA3D, At Baseline: number analyzed (Participants) | 4
  Gene: SEMA3D, At Baseline | 45.814 (5.7690)
  Gene: SEMA3D, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3D, Change at Week 16 | -1.638 (0.6445)
  Gene: SEMA3E, At Baseline: number analyzed (Participants) | 6
  Gene: SEMA3E, At Baseline | 43.005 (1.6275)
  Gene: SEMA3E, Change at Week 16: number analyzed (Participants) | 4
  Gene: SEMA3E, Change at Week 16 | -3.132 (2.4180)
  Gene: SEMA3F, At Baseline: number analyzed (Participants) | 4
  Gene: SEMA3F, At Baseline | 54.979 (15.1825)
  Gene: SEMA3F, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3F, Change at Week 16 | -3.556 (1.1758)
  Gene: SEMA3G, At Baseline: number analyzed (Participants) | 24
  Gene: SEMA3G, At Baseline | 44.464 (8.4848)
  Gene: SEMA3G, Change at Week 16: number analyzed (Participants) | 14
  Gene: SEMA3G, Change at Week 16 | -2.124 (1.5203)
  Gene: PHIP, At Baseline: number analyzed (Participants) | 16
  Gene: PHIP, At Baseline | 40.808 (10.0222)
  Gene: PHIP, Change at Week 16: number analyzed (Participants) | 13
  Gene: PHIP, Change at Week 16 | -2.120 (1.0108)
  Gene: SIM1, At Baseline: number analyzed (Participants) | 20
  Gene: SIM1, At Baseline | 47.729 (9.7294)
  Gene: SIM1, Change at Week 16: number analyzed (Participants) | 16
  Gene: SIM1, Change at Week 16 | -1.698 (1.8931)
  Gene: MAGEL2, At Baseline: number analyzed (Participants) | 10
  Gene: MAGEL2, At Baseline | 42.047 (8.2605)
  Gene: MAGEL2, Change at Week 16: number analyzed (Participants) | 7
  Gene: MAGEL2, Change at Week 16 | -1.637 (1.3549)
  Gene: CREBBP, At Baseline: number analyzed (Participants) | 1
  Gene: CREBBP, At Baseline | 47.490
  Gene: CREBBP, Change at Week 16: number analyzed (Participants) | 1
  Gene: CREBBP, Change at Week 16 | 0.165
  Gene: DNMT3A, At Baseline: number analyzed (Participants) | 1
  Gene: DNMT3A, At Baseline | 44.138
  Gene: DNMT3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: DNMT3A, Change at Week 16 | -1.080
  Gene: HTR2C, At Baseline: number analyzed (Participants) | 3
  Gene: HTR2C, At Baseline | 52.105 (3.0212)
  Gene: HTR2C, Change at Week 16: number analyzed (Participants) | 1
  Gene: HTR2C, Change at Week 16 | -1.381
  Gene: KSR2, At Baseline: number analyzed (Participants) | 11
  Gene: KSR2, At Baseline | 47.624 (11.4457)
  Gene: KSR2, Change at Week 16: number analyzed (Participants) | 8
  Gene: KSR2, Change at Week 16 | -1.073 (1.4410)
  Gene: MRAP2, At Baseline: number analyzed (Participants) | 1
  Gene: MRAP2, At Baseline | 58.100
  Gene: MRAP2, Change at Week 16: number analyzed (Participants) | 1
  Gene: MRAP2, Change at Week 16 | -1.470
  Gene: RPGRIP1L, At Baseline: number analyzed (Participants) | 3
  Gene: RPGRIP1L, At Baseline | 43.442 (2.6778)
  Gene: RPGRIP1L, Change at Week 16: number analyzed (Participants) | 1
  Gene: RPGRIP1L, Change at Week 16 | -3.603
  Gene: TBX3, At Baseline: number analyzed (Participants) | 5
  Gene: TBX3, At Baseline | 40.170 (10.5867)
  Gene: TBX3, Change at Week 16: number analyzed (Participants) | 3
  Gene: TBX3, Change at Week 16 | -1.951 (1.3582)
  Gene: TRPC5, At Baseline: number analyzed (Participants) | 3
  Gene: TRPC5, At Baseline | 49.974 (24.5155)
  Gene: TRPC5, Change at Week 16: number analyzed (Participants) | 2
  Gene: TRPC5, Change at Week 16 | 0.161 (1.2979)

3. Secondary Outcome: Mean Change in BMI From Baseline to the End of Stage 1 in Participants ≥18 Years Old, Per Genotype
Description: BMI was calculated using participant's weight and height assessments, using the following formula: BMI = kg/m^2 Data are provided for overall and according to participants with specified primary gene.
  Baseline was defined as the last available measurement taken prior to the start of treatment Stage 1 administration.
Time Frame: Baseline, Week 16
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Kg/m^2
Groups:
- Stage 1: Setmelanotide (Open-Label): Participants received once daily SC injection of setmelanotide from Day 1 to Week 16 in an open-label treatment stage (Stage 1). Participants ≥12 years of age started on setmelanotide 2.0 mg once daily for approximately 2 weeks, then increased to 3.0 mg once daily.
Arm/Group | Stage 1: Setmelanotide (Open-Label)
Number analyzed (Participants) | 109
Kg/m^2
  Overall: At Baseline | 48.464 (8.0877)
  Overall: Change at Week 16: number analyzed (Participants) | 69
  Overall: Change at Week 16 | -1.872 (1.8963)
  Gene: NRP2, At Baseline: number analyzed (Participants) | 2
  Gene: NRP2, At Baseline | 51.640 (8.5762)
  Gene: NRP2, Change at Week 16: number analyzed (Participants) | 2
  Gene: NRP2, Change at Week 16 | -0.783 (1.0489)
  Gene: PLXNA1, At Baseline: number analyzed (Participants) | 5
  Gene: PLXNA1, At Baseline | 46.959 (6.2279)
  Gene: PLXNA1, Change at Week 16: number analyzed (Participants) | 3
  Gene: PLXNA1, Change at Week 16 | -0.678 (0.8796)
  Gene: PLXNA2, At Baseline: number analyzed (Participants) | 7
  Gene: PLXNA2, At Baseline | 50.335 (12.3004)
  Gene: PLXNA2, Change at Week 16: number analyzed (Participants) | 4
  Gene: PLXNA2, Change at Week 16 | -2.324 (0.6565)
  Gene: PLXNA3, At Baseline: number analyzed (Participants) | 1
  Gene: PLXNA3, At Baseline | 40.801
  Gene: PLXNA3, Change at Week 16: number analyzed (Participants) | 1
  Gene: PLXNA3, Change at Week 16 | -3.698
  Gene: PLXNA4, At Baseline: number analyzed (Participants) | 17
  Gene: PLXNA4, At Baseline | 48.420 (7.4340)
  Gene: PLXNA4, Change at Week 16: number analyzed (Participants) | 11
  Gene: PLXNA4, Change at Week 16 | -2.532 (3.1514)
  Gene: SEMA3A, At Baseline: number analyzed (Participants) | 1
  Gene: SEMA3A, At Baseline | 47.366
  Gene: SEMA3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3A, Change at Week 16 | -2.513
  Gene: SEMA3B, At Baseline: number analyzed (Participants) | 1
  Gene: SEMA3B, At Baseline | 43.320
  Gene: SEMA3B, Change at Week 16: number analyzed (Participants) | 0
  Gene: SEMA3D, At Baseline: number analyzed (Participants) | 3
  Gene: SEMA3D, At Baseline | 47.296 (6.0613)
  Gene: SEMA3D, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3D, Change at Week 16 | -1.638 (0.6445)
  Gene: SEMA3E, At Baseline: number analyzed (Participants) | 2
  Gene: SEMA3E, At Baseline | 42.004 (1.1954)
  Gene: SEMA3E, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3E, Change at Week 16 | -4.716 (0.0565)
  Gene: SEMA3F, At Baseline: number analyzed (Participants) | 2
  Gene: SEMA3F, At Baseline | 64.964 (9.9946)
  Gene: SEMA3F, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3F, Change at Week 16 | -4.388
  Gene: SEMA3G, At Baseline: number analyzed (Participants) | 18
  Gene: SEMA3G, At Baseline | 46.762 (6.5047)
  Gene: SEMA3G, Change at Week 16: number analyzed (Participants) | 9
  Gene: SEMA3G, Change at Week 16 | -2.302 (1.6478)
  Gene: PHIP, At Baseline: number analyzed (Participants) | 10
  Gene: PHIP, At Baseline | 45.343 (7.0089)
  Gene: PHIP, Change at Week 16: number analyzed (Participants) | 7
  Gene: PHIP, Change at Week 16 | -2.110 (1.1464)
  Gene: SIM1, At Baseline: number analyzed (Participants) | 13
  Gene: SIM1, At Baseline | 50.790 (8.9593)
  Gene: SIM1, Change at Week 16: number analyzed (Participants) | 10
  Gene: SIM1, Change at Week 16 | -1.465 (1.7916)
  Gene: MAGEL2, At Baseline: number analyzed (Participants) | 7
  Gene: MAGEL2, At Baseline | 46.198 (5.0997)
  Gene: MAGEL2, Change at Week 16: number analyzed (Participants) | 4
  Gene: MAGEL2, Change at Week 16 | -1.191 (1.0137)
  Gene: CREBBP, At Baseline: number analyzed (Participants) | 1
  Gene: CREBBP, At Baseline | 47.490
  Gene: CREBBP, Change at Week 16: number analyzed (Participants) | 1
  Gene: CREBBP, Change at Week 16 | 0.165
  Gene: DNMT3A, At Baseline: number analyzed (Participants) | 1
  Gene: DNMT3A, At Baseline | 44.138
  Gene: DNMT3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: DNMT3A, Change at Week 16 | -1.080
  Gene: HTR2C, At Baseline: number analyzed (Participants) | 3
  Gene: HTR2C, At Baseline | 52.105 (3.0212)
  Gene: HTR2C, Change at Week 16: number analyzed (Participants) | 1
  Gene: HTR2C, Change at Week 16 | -1.381
  Gene: KSR2, At Baseline: number analyzed (Participants) | 8
  Gene: KSR2, At Baseline | 51.397 (9.2011)
  Gene: KSR2, Change at Week 16: number analyzed (Participants) | 5
  Gene: KSR2, Change at Week 16 | -0.792 (1.5759)
  Gene: RPGRIP1L, At Baseline: number analyzed (Participants) | 3
  Gene: RPGRIP1L, At Baseline | 43.442 (2.6778)
  Gene: RPGRIP1L, Change at Week 16: number analyzed (Participants) | 1
  Gene: RPGRIP1L, Change at Week 16 | -3.603
  Gene: TBX3, At Baseline: number analyzed (Participants) | 2
  Gene: TBX3, At Baseline | 44.494 (4.3444)
  Gene: TBX3, Change at Week 16: number analyzed (Participants) | 1
  Gene: TBX3, Change at Week 16 | -0.705
  Gene: TRPC5, At Baseline: number analyzed (Participants) | 2
  Gene: TRPC5, At Baseline | 62.246 (17.2758)
  Gene: TRPC5, Change at Week 16: number analyzed (Participants) | 2
  Gene: TRPC5, Change at Week 16 | 0.161 (1.2979)

4. Secondary Outcome: Percent Change in BMI From Baseline to the End of Stage 1 in All Participants, Per Genotype
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Stage 1: Setmelanotide (Open-Label)
Number analyzed (Participants) | 112
percent change
  Overall: Change at Week 16 | -4.62 (4.394)
  Gene: NRP1, Change at Week 16: number analyzed (Participants) | 2
  Gene: NRP1, Change at Week 16 | 0.57 (3.329)
  Gene: PLXNA1, Change at Week 16: number analyzed (Participants) | 5
  Gene: PLXNA1, Change at Week 16 | -4.00 (4.296)
  Gene: NRP2, Change at Week 16: number analyzed (Participants) | 3
  Gene: NRP2, Change at Week 16 | -2.33 (2.105)
  Gene: PLXNA2, Change at Week 16: number analyzed (Participants) | 6
  Gene: PLXNA2, Change at Week 16 | -4.90 (3.909)
  Gene: PLXNA3, Change at Week 16: number analyzed (Participants) | 2
  Gene: PLXNA3, Change at Week 16 | -8.95 (0.156)
  Gene: PLXNA4, Change at Week 16: number analyzed (Participants) | 14
  Gene: PLXNA4, Change at Week 16 | -5.00 (6.577)
  Gene: SEMA3A, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3A, Change at Week 16 | -5.39 (0.123)
  Gene: SEMA3B, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3B, Change at Week 16 | -6.79
  Gene: SEMA3C, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3C, Change at Week 16 | -4.91
  Gene: SEMA3D, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3D, Change at Week 16 | -3.57 (1.960)
  Gene: SEMA3E, Change at Week 16: number analyzed (Participants) | 4
  Gene: SEMA3E, Change at Week 16 | -7.39 (5.752)
  Gene: SEMA3F, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3F, Change at Week 16 | -7.66 (0.119)
  Gene: SEMA3G, Change at Week 16: number analyzed (Participants) | 14
  Gene: SEMA3G, Change at Week 16 | -5.09 (3.284)
  Gene: PHIP, Change at Week 16: number analyzed (Participants) | 13
  Gene: PHIP, Change at Week 16 | -6.12 (3.623)
  Gene: SIM1, Change at Week 16: number analyzed (Participants) | 16
  Gene: SIM1, Change at Week 16 | -4.02 (5.310)
  Gene: MAGEL2, Change at Week 16: number analyzed (Participants) | 7
  Gene: MAGEL2, Change at Week 16 | -4.60 (4.288)
  Gene: CREBBP, Change at Week 16: number analyzed (Participants) | 1
  Gene: CREBBP, Change at Week 16 | 0.35
  Gene: DNMT3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: DNMT3A, Change at Week 16 | -2.45
  Gene: HTR2C, Change at Week 16: number analyzed (Participants) | 1
  Gene: HTR2C, Change at Week 16 | -2.49
  Gene: KSR2, Change at Week 16: number analyzed (Participants) | 8
  Gene: KSR2, Change at Week 16 | -2.15 (2.928)
  Gene: MRAP2, Change at Week 16: number analyzed (Participants) | 1
  Gene: MRAP2, Change at Week 16 | -2.53
  Gene: RPGRIP1L, Change at Week 16: number analyzed (Participants) | 1
  Gene: RPGRIP1L, Change at Week 16 | -8.64
  Gene: TBX3, Change at Week 16: number analyzed (Participants) | 3
  Gene: TBX3, Change at Week 16 | -6.41 (5.011)
  Gene: TRPC5, Change at Week 16: number analyzed (Participants) | 2
  Gene: TRPC5, Change at Week 16 | -0.03 (2.094)

5. Secondary Outcome: Percent Change in BMI From Baseline to the End of Stage 1 in Participants ≥18 Years Old, Per Genotype
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Stage 1: Setmelanotide (Open-Label)
Number analyzed (Participants) | 69
percent change
  Overall: Change at Week 16 | -3.95 (4.057)
  Gene: NRP2, Change at Week 16: number analyzed (Participants) | 2
  Gene: NRP2, Change at Week 16 | -1.37 (1.804)
  Gene: PLXNA1, Change at Week 16: number analyzed (Participants) | 3
  Gene: PLXNA1, Change at Week 16 | -1.22 (1.576)
  Gene: PLXNA2, Change at Week 16: number analyzed (Participants) | 4
  Gene: PLXNA2, Change at Week 16 | -4.69 (0.913)
  Gene: PLXNA3, Change at Week 16: number analyzed (Participants) | 1
  Gene: PLXNA3, Change at Week 16 | -9.06
  Gene: PLXNA4, Change at Week 16: number analyzed (Participants) | 11
  Gene: PLXNA4, Change at Week 16 | -5.34 (6.682)
  Gene: SEMA3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3A, Change at Week 16 | -5.31
  Gene: SEMA3D, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3D, Change at Week 16 | -3.57 (1.960)
  Gene: SEMA3E, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3E, Change at Week 16 | -11.23 (0.185)
  Gene: SEMA3F, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3F, Change at Week 16 | -7.58
  Gene: SEMA3G, Change at Week 16: number analyzed (Participants) | 9
  Gene: SEMA3G, Change at Week 16 | -4.80 (2.810)
  Gene: PHIP, Change at Week 16: number analyzed (Participants) | 7
  Gene: PHIP, Change at Week 16 | -5.11 (2.770)
  Gene: SIM1, Change at Week 16: number analyzed (Participants) | 10
  Gene: SIM1, Change at Week 16 | -2.63 (3.720)
  Gene: MAGEL2, Change at Week 16: number analyzed (Participants) | 4
  Gene: MAGEL2, Change at Week 16 | -2.67 (2.227)
  Gene: CREBBP, Change at Week 16: number analyzed (Participants) | 1
  Gene: CREBBP, Change at Week 16 | 0.35
  Gene: DNMT3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: DNMT3A, Change at Week 16 | -2.45
  Gene: HTR2C, Change at Week 16: number analyzed (Participants) | 1
  Gene: HTR2C, Change at Week 16 | -2.49
  Gene: KSR2, Change at Week 16: number analyzed (Participants) | 5
  Gene: KSR2, Change at Week 16 | -1.23 (3.189)
  Gene: RPGRIP1L, Change at Week 16: number analyzed (Participants) | 1
  Gene: RPGRIP1L, Change at Week 16 | -8.64
  Gene: TBX3, Change at Week 16: number analyzed (Participants) | 1
  Gene: TBX3, Change at Week 16 | -1.70
  Gene: TRPC5, Change at Week 16: number analyzed (Participants) | 2
  Gene: TRPC5, Change at Week 16 | -0.03 (2.094)

6. Secondary Outcome: Mean Change in Body Weight From Baseline to the End of Stage 1 in Participants ≥18 Years Old, Per Genotype
Description: Data are provided for overall and according to participants with specified primary gene.
  Baseline was defined as the last available measurement taken prior to the start of treatment Stage 1 administration.
Time Frame: Baseline, Week 16
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Stage 1: Setmelanotide (Open-Label)
Number analyzed (Participants) | 109
Kg
  Overall, At Baseline | 136.01 (29.815)
  Overall: Change at Week 16: number analyzed (Participants) | 69
  Overall: Change at Week 16 | -5.33 (5.315)
  Gene: NRP2, At Baseline: number analyzed (Participants) | 2
  Gene: NRP2, At Baseline | 147.35 (2.098)
  Gene: NRP2, Change at Week 16: number analyzed (Participants) | 2
  Gene: NRP2, Change at Week 16 | -2.03 (2.687)
  Gene: PLXNA1, At Baseline: number analyzed (Participants) | 5
  Gene: PLXNA1, At Baseline | 145.30 (33.751)
  Gene: PLXNA1, Change at Week 16: number analyzed (Participants) | 3
  Gene: PLXNA1, Change at Week 16 | -2.33 (3.144)
  Gene: PLXNA2, At Baseline: number analyzed (Participants) | 7
  Gene: PLXNA2, At Baseline | 137.94 (37.878)
  Gene: PLXNA2, Change at Week 16: number analyzed (Participants) | 4
  Gene: PLXNA2, Change at Week 16 | -6.50 (2.234)
  Gene: PLXNA3, At Baseline: number analyzed (Participants) | 1
  Gene: PLXNA3, At Baseline | 89.73
  Gene: PLXNA3, Change at Week 16: number analyzed (Participants) | 1
  Gene: PLXNA3, Change at Week 16 | -8.13
  Gene: PLXNA4, At Baseline: number analyzed (Participants) | 17
  Gene: PLXNA4, At Baseline | 135.87 (24.052)
  Gene: PLXNA4, Change at Week 16: number analyzed (Participants) | 11
  Gene: PLXNA4, Change at Week 16 | -7.55 (8.772)
  Gene: SEMA3A, At Baseline: number analyzed (Participants) | 1
  Gene: SEMA3A, At Baseline | 157.07
  Gene: SEMA3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3A, Change at Week 16 | -8.33
  Gene: SEMA3B, At Baseline: number analyzed (Participants) | 1
  Gene: SEMA3B, At Baseline | 97.60
  Gene: SEMA3B, Change at Week 16: number analyzed (Participants) | 0
  Gene: SEMA3D, At Baseline: number analyzed (Participants) | 3
  Gene: SEMA3D, At Baseline | 128.09 (49.981)
  Gene: SEMA3D, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3D, Change at Week 16 | -4.48 (0.589)
  Gene: SEMA3E, At Baseline: number analyzed (Participants) | 2
  Gene: SEMA3E, At Baseline | 115.77 (19.328)
  Gene: SEMA3E, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3E, Change at Week 16 | -12.98 (1.956)
  Gene: SEMA3F, At Baseline: number analyzed (Participants) | 2
  Gene: SEMA3F, At Baseline | 176.65 (10.960)
  Gene: SEMA3F, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3F, Change at Week 16 | -12.80
  Gene: SEMA3G, At Baseline: number analyzed (Participants) | 18
  Gene: SEMA3G, At Baseline | 129.41 (21.874)
  Gene: SEMA3G, Change at Week 16: number analyzed (Participants) | 9
  Gene: SEMA3G, Change at Week 16 | -6.59 (4.622)
  Gene: PHIP, At Baseline: number analyzed (Participants) | 10
  Gene: PHIP, At Baseline | 134.11 (36.996)
  Gene: PHIP, Change at Week 16: number analyzed (Participants) | 7
  Gene: PHIP, Change at Week 16 | -5.77 (3.504)
  Gene: SIM1, At Baseline: number analyzed (Participants) | 13
  Gene: SIM1, At Baseline | 141.25 (35.591)
  Gene: SIM1, Change at Week 16: number analyzed (Participants) | 10
  Gene: SIM1, Change at Week 16 | -4.13 (4.720)
  Gene: MAGEL2, At Baseline: number analyzed (Participants) | 7
  Gene: MAGEL2, At Baseline | 134.41 (20.544)
  Gene: MAGEL2, Change at Week 16: number analyzed (Participants) | 4
  Gene: MAGEL2, Change at Week 16 | -3.88 (3.681)
  Gene: CREBBP, At Baseline: number analyzed (Participants) | 1
  Gene: CREBBP, At Baseline | 103.60
  Gene: CREBBP, Change at Week 16: number analyzed (Participants) | 1
  Gene: CREBBP, Change at Week 16 | 0.36
  Gene: DNMT3A, At Baseline: number analyzed (Participants) | 1
  Gene: DNMT3A, At Baseline | 129.37
  Gene: DNMT3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: DNMT3A, Change at Week 16 | -3.17
  Gene: HTR2C, At Baseline: number analyzed (Participants) | 3
  Gene: HTR2C, At Baseline | 126.23 (9.780)
  Gene: HTR2C, Change at Week 16: number analyzed (Participants) | 1
  Gene: HTR2C, Change at Week 16 | -3.40
  Gene: KSR2, At Baseline: number analyzed (Participants) | 8
  Gene: KSR2, At Baseline | 150.16 (19.630)
  Gene: KSR2, Change at Week 16: number analyzed (Participants) | 5
  Gene: KSR2, Change at Week 16 | -2.13 (4.721)
  Gene: RPGRIP1L, At Baseline: number analyzed (Participants) | 3
  Gene: RPGRIP1L, At Baseline | 103.47 (11.193)
  Gene: RPGRIP1L, Change at Week 16: number analyzed (Participants) | 1
  Gene: RPGRIP1L, Change at Week 16 | -8.63
  Gene: TBX3, At Baseline: number analyzed (Participants) | 2
  Gene: TBX3, At Baseline | 119.00 (11.644)
  Gene: TBX3, Change at Week 16: number analyzed (Participants) | 1
  Gene: TBX3, Change at Week 16 | -2.17
  Gene: TRPC5, At Baseline: number analyzed (Participants) | 2
  Gene: TRPC5, At Baseline | 203.00 (25.173)
  Gene: TRPC5, Change at Week 16: number analyzed (Participants) | 2
  Gene: TRPC5, Change at Week 16 | 0.20 (4.243)

7. Secondary Outcome: Percent Change in Body Weight From Baseline to the End of Stage 1 in Participants ≥18 Years Old, Per Genotype
Description: as for outcome 6
Time Frame: Baseline, Week 16
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Stage 1: Setmelanotide (Open-Label)
Number analyzed (Participants) | 69
percent change
  Overall: Change at Week 16 | -3.94 (4.052)
  Gene: NRP2, Change at Week 16: number analyzed (Participants) | 2
  Gene: NRP2, Change at Week 16 | -1.37 (1.804)
  Gene: PLXNA1, Change at Week 16: number analyzed (Participants) | 3
  Gene: PLXNA1, Change at Week 16 | -1.22 (1.576)
  Gene: PLXNA2, Change at Week 16: number analyzed (Participants) | 4
  Gene: PLXNA2, Change at Week 16 | -4.69 (0.913)
  Gene: PLXNA3, Change at Week 16: number analyzed (Participants) | 1
  Gene: PLXNA3, Change at Week 16 | -9.06
  Gene: PLXNA4, Change at Week 16: number analyzed (Participants) | 11
  Gene: PLXNA4, Change at Week 16 | -5.34 (6.682)
  Gene: SEMA3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3A, Change at Week 16 | -5.31
  Gene: SEMA3D, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3D, Change at Week 16 | -3.57 (1.960)
  Gene: SEMA3E, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3E, Change at Week 16 | -11.23 (0.185)
  Gene: SEMA3F, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3F, Change at Week 16 | -7.58
  Gene: SEMA3G, Change at Week 16: number analyzed (Participants) | 9
  Gene: SEMA3G, Change at Week 16 | -4.80 (2.810)
  Gene: PHIP, Change at Week 16: number analyzed (Participants) | 7
  Gene: PHIP, Change at Week 16 | -5.00 (2.749)
  Gene: SIM1, Change at Week 16: number analyzed (Participants) | 10
  Gene: SIM1, Change at Week 16 | -2.63 (3.720)
  Gene: MAGEL2, Change at Week 16: number analyzed (Participants) | 4
  Gene: MAGEL2, Change at Week 16 | -2.67 (2.227)
  Gene: CREBBP, Change at Week 16: number analyzed (Participants) | 1
  Gene: CREBBP, Change at Week 16 | 0.35
  Gene: DNMT3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: DNMT3A, Change at Week 16 | -2.45
  Gene: HTR2C, Change at Week 16: number analyzed (Participants) | 1
  Gene: HTR2C, Change at Week 16 | -2.49
  Gene: KSR2, Change at Week 16: number analyzed (Participants) | 5
  Gene: KSR2, Change at Week 16 | -1.23 (3.189)
  Gene: RPGRIP1L, Change at Week 16: number analyzed (Participants) | 1
  Gene: RPGRIP1L, Change at Week 16 | -8.64
  Gene: TBX3, Change at Week 16: number analyzed (Participants) | 1
  Gene: TBX3, Change at Week 16 | -1.70
  Gene: TRPC5, Change at Week 16: number analyzed (Participants) | 2
  Gene: TRPC5, Change at Week 16 | -0.03 (2.094)

8. Secondary Outcome: Mean Change in BMI Z-score From Baseline to the End of Stage 1 in Participants <18 Years Old, Per Genotype
Description: BMI was calculated using participant's weight and height assessments, using the following formula: BMI = kg/m^2. The BMI Z-score indicated the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). A decrease of BMI Z-score indicates a reduction in BMI from Baseline whereas an increase of BMI-Z score indicates an increase in BMI from Baseline.
  Baseline was defined as the last available measurement taken prior to the start of treatment Stage 1 administration.
Time Frame: Baseline, Week 16
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Stage 1: Setmelanotide (Open-Label): Participants received once daily SC injection of setmelanotide from Day 1 to Week 16 in an open-label treatment stage (Stage 1). Participants ≥12 years of age started on setmelanotide 2.0 mg once daily for approximately 2 weeks, then increased to 3.0 mg once daily. Participants <12 years of age started on setmelanotide 1.0 mg once daily for approximately 1 week, then increased to 2.0 mg once daily for approximately 1 week, then increased to 3 mg once daily.
Arm/Group | Stage 1: Setmelanotide (Open-Label)
Number analyzed (Participants) | 55
z-score
  Overall, At Baseline | 2.649 (0.3708)
  Overall: Change at Week 16: number analyzed (Participants) | 43
  Overall: Change at Week 16 | -0.126 (0.1425)
  Gene: NRP1, At Baseline: number analyzed (Participants) | 2
  Gene: NRP1, At Baseline | 2.919 (0.0848)
  Gene: NRP1, Change at Week 16: number analyzed (Participants) | 2
  Gene: NRP1, Change at Week 16 | -0.000 (0.0124)
  Gene: NRP2, At Baseline: number analyzed (Participants) | 1
  Gene: NRP2, At Baseline | 2.386
  Gene: NRP2, Change at Week 16: number analyzed (Participants) | 1
  Gene: NRP2, Change at Week 16 | -0.086
  Gene: PLXNA1, At Baseline: number analyzed (Participants) | 3
  Gene: PLXNA1, At Baseline | 2.729 (0.1250)
  Gene: PLXNA1, Change at Week 16: number analyzed (Participants) | 2
  Gene: PLXNA1, Change at Week 16 | -0.112 (0.0671)
  Gene: PLXNA2, At Baseline: number analyzed (Participants) | 2
  Gene: PLXNA2, At Baseline | 2.955 (0.0601)
  Gene: PLXNA2, Change at Week 16: number analyzed (Participants) | 2
  Gene: PLXNA2, Change at Week 16 | -0.043 (0.0707)
  Gene: PLXNA3, At Baseline: number analyzed (Participants) | 2
  Gene: PLXNA3, At Baseline | 2.485 (0.4970)
  Gene: PLXNA3, Change at Week 16: number analyzed (Participants) | 1
  Gene: PLXNA3, Change at Week 16 | -0.234
  Gene: PLXNA4, At Baseline: number analyzed (Participants) | 3
  Gene: PLXNA4, At Baseline | 2.693 (0.3653)
  Gene: PLXNA4, Change at Week 16: number analyzed (Participants) | 3
  Gene: PLXNA4, Change at Week 16 | -0.063 (0.1110)
  Gene: SEMA3A, At Baseline: number analyzed (Participants) | 2
  Gene: SEMA3A, At Baseline | 2.498 (0.2057)
  Gene: SEMA3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3A, Change at Week 16 | -0.078
  Gene: SEMA3B, At Baseline: number analyzed (Participants) | 2
  Gene: SEMA3B, At Baseline | 2.595 (0.5201)
  Gene: SEMA3B, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3B, Change at Week 16 | -0.140
  Gene: SEMA3C, At Baseline: number analyzed (Participants) | 1
  Gene: SEMA3C, At Baseline | 2.828
  Gene: SEMA3C, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3C, Change at Week 16 | -0.037
  Gene: SEMA3D, At Baseline: number analyzed (Participants) | 1
  Gene: SEMA3D, At Baseline | 2.454
  Gene: SEMA3D, Change at Week 16: number analyzed (Participants) | 0
  Gene: SEMA3E, At Baseline: number analyzed (Participants) | 4
  Gene: SEMA3E, At Baseline | 2.913 (0.4705)
  Gene: SEMA3E, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3E, Change at Week 16 | -0.053 (0.0808)
  Gene: SEMA3F, At Baseline: number analyzed (Participants) | 2
  Gene: SEMA3F, At Baseline | 2.847 (0.5676)
  Gene: SEMA3F, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3F, Change at Week 16 | -0.192
  Gene: SEMA3G, At Baseline: number analyzed (Participants) | 6
  Gene: SEMA3G, At Baseline | 2.826 (0.4890)
  Gene: SEMA3G, Change at Week 16: number analyzed (Participants) | 5
  Gene: SEMA3G, Change at Week 16 | -0.115 (0.1020)
  Gene: PHIP, At Baseline: number analyzed (Participants) | 6
  Gene: PHIP, At Baseline | 2.457 (0.4515)
  Gene: PHIP, Change at Week 16: number analyzed (Participants) | 6
  Gene: PHIP, Change at Week 16 | -0.201 (0.1923)
  Gene: SIM1, At Baseline: number analyzed (Participants) | 7
  Gene: SIM1, At Baseline | 2.510 (0.3107)
  Gene: SIM1, Change at Week 16: number analyzed (Participants) | 6
  Gene: SIM1, Change at Week 16 | -0.182 (0.2355)
  Gene: MAGEL2, At Baseline: number analyzed (Participants) | 3
  Gene: MAGEL2, At Baseline | 2.503 (0.3034)
  Gene: MAGEL2, Change at Week 16: number analyzed (Participants) | 3
  Gene: MAGEL2, Change at Week 16 | -0.184 (0.1615)
  Gene: MRAP2, At Baseline: number analyzed (Participants) | 1
  Gene: MRAP2, At Baseline | 2.738
  Gene: MRAP2, Change at Week 16: number analyzed (Participants) | 1
  Gene: MRAP2, Change at Week 16 | -0.019
  Gene: KSR2, At Baseline: number analyzed (Participants) | 3
  Gene: KSR2, At Baseline | 2.831 (0.2260)
  Gene: KSR2, Change at Week 16: number analyzed (Participants) | 3
  Gene: KSR2, Change at Week 16 | -0.037 (0.0131)
  Gene: TBX3, At Baseline: number analyzed (Participants) | 3
  Gene: TBX3, At Baseline | 2.471 (0.4419)
  Gene: TBX3, Change at Week 16: number analyzed (Participants) | 2
  Gene: TBX3, Change at Week 16 | -0.254 (0.1661)
  Gene: TRPC5, At Baseline: number analyzed (Participants) | 1
  Gene: TRPC5, At Baseline | 2.078
  Gene: TRPC5, Change at Week 16: number analyzed (Participants) | 0

9. Secondary Outcome: Percent Change in the Weekly Average of the Daily Maximal Hunger Score From Baseline to the End of Stage 1 in Participants ≥12 Years Old, Per Genotype
Description: Daily Hunger Questionnaire for participants ≥12 years of age is self-administered questionnaire and comprises three items. For the assessment of this endpoint, maximal hunger was corresponding to the following question: In the last 24 hours, how hungry did you feel when you were the most hungry? The response was scored separately and averaged on weekly basis. Participants rated their hunger on an 11-point numeric rating scale ranging from 0 to 10 (0 = not hungry at all, and 10 = hungriest possible).
  Weekly average at Week 16 was defined as average of the available score values within 7 days in Week 16.
  Baseline was defined as the average of the available score values within 7 days before or on the stage 1 open-label treatment.
  Results are reported by overall participant results and by specific gene cohort.
Time Frame: Baseline, Week 16
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Stage 1: Setmelanotide (Open-Label)
Number analyzed (Participants) | 139
percent change
  Overall: Change at Week 16: number analyzed (Participants) | 78
  Overall: Change at Week 16 | -31.13 (63.273)
  Gene: NRP2, Change at Week 16: number analyzed (Participants) | 2
  Gene: NRP2, Change at Week 16 | -39.63 (1.203)
  Gene: PLXNA1, Change at Week 16: number analyzed (Participants) | 3
  Gene: PLXNA1, Change at Week 16 | -21.04 (10.064)
  Gene: PLXNA2, Change at Week 16: number analyzed (Participants) | 5
  Gene: PLXNA2, Change at Week 16 | -44.12 (37.973)
  Gene: PLXNA3, Change at Week 16: number analyzed (Participants) | 2
  Gene: PLXNA3, Change at Week 16 | -49.25 (4.785)
  Gene: PLXNA4, Change at Week 16: number analyzed (Participants) | 9
  Gene: PLXNA4, Change at Week 16 | -54.61 (31.759)
  Gene: SEMA3A, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3A, Change at Week 16 | -15.35 (5.880)
  Gene: SEMA3B, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3B, Change at Week 16 | -15.79
  Gene: SEMA3C, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3C, Change at Week 16 | 0.00
  Gene: SEMA3D, Change at Week 16: number analyzed (Participants) | 1
  Gene: SEMA3D, Change at Week 16 | 36.36
  Gene: SEMA3E, Change at Week 16: number analyzed (Participants) | 3
  Gene: SEMA3E, Change at Week 16 | -37.37 (23.609)
  Gene: SEMA3F, Change at Week 16: number analyzed (Participants) | 2
  Gene: SEMA3F, Change at Week 16 | -48.16 (24.821)
  Gene: SEMA3G, Change at Week 16: number analyzed (Participants) | 7
  Gene: SEMA3G, Change at Week 16 | 38.70 (176.373)
  Gene: PHIP, Change at Week 16: number analyzed (Participants) | 8
  Gene: PHIP, Change at Week 16 | -56.87 (19.460)
  Gene: SIM1, Change at Week 16: number analyzed (Participants) | 14
  Gene: SIM1, Change at Week 16 | -25.60 (51.690)
  Gene: MAGEL2, Change at Week 16: number analyzed (Participants) | 6
  Gene: MAGEL2, Change at Week 16 | -39.44 (30.215)
  Gene: CREBBP, Change at Week 16: number analyzed (Participants) | 0
  Gene: DNMT3A, Change at Week 16: number analyzed (Participants) | 1
  Gene: DNMT3A, Change at Week 16 | -23.00
  Gene: HTR2C, Change at Week 16: number analyzed (Participants) | 1
  Gene: HTR2C, Change at Week 16 | -37.29
  Gene: KSR2, Change at Week 16: number analyzed (Participants) | 4
  Gene: KSR2, Change at Week 16 | -42.17 (30.842)
  Gene: MRAP2, Change at Week 16: number analyzed (Participants) | 1
  Gene: MRAP2, Change at Week 16 | -47.83
  Gene: RPGRIP1L, Change at Week 16: number analyzed (Participants) | 1
  Gene: RPGRIP1L, Change at Week 16 | -100.00
  Gene: TBX3, Change at Week 16: number analyzed (Participants) | 2
  Gene: TBX3, Change at Week 16 | -33.67 (2.720)
  Gene: TRPC5, Change at Week 16: number analyzed (Participants) | 2
  Gene: TRPC5, Change at Week 16 | -16.82 (28.427)

10. Secondary Outcome: Number of Participants ≥12 Years Old, Who Achieved a ≥2 Point Reduction From Baseline to the End of Stage 1 in the Weekly Average of the Daily Maximal Hunger Score, Per Genotype
Description: as for outcome 9
Time Frame: Baseline, Week 16
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Setmelanotide (Open-Label)
Number analyzed (Participants) | 141
Participants
  Overall | 49
  Gene: NRP2: number analyzed (Participants) | 3
  Gene: NRP2 | 2
  Gene: PLXNA1: number analyzed (Participants) | 8
  Gene: PLXNA1 | 1
  Gene: PLXNA2: number analyzed (Participants) | 8
  Gene: PLXNA2 | 3
  Gene: PLXNA3: number analyzed (Participants) | 2
  Gene: PLXNA3 | 2
  Gene: PLXNA4: number analyzed (Participants) | 19
  Gene: PLXNA4 | 6
  Gene: SEMA3A: number analyzed (Participants) | 3
  Gene: SEMA3A | 0
  Gene: SEMA3B: number analyzed (Participants) | 2
  Gene: SEMA3B | 0
  Gene: SEMA3C: number analyzed (Participants) | 1
  Gene: SEMA3C | 0
  Gene: SEMA3D: number analyzed (Participants) | 4
  Gene: SEMA3D | 0
  Gene: SEMA3E: number analyzed (Participants) | 5
  Gene: SEMA3E | 2
  Gene: SEMA3F: number analyzed (Participants) | 4
  Gene: SEMA3F | 2
  Gene: SEMA3G: number analyzed (Participants) | 18
  Gene: SEMA3G | 4
  Gene: PHIP: number analyzed (Participants) | 12
  Gene: PHIP | 7
  Gene: SIM1: number analyzed (Participants) | 20
  Gene: SIM1 | 7
  Gene: MAGEL2: number analyzed (Participants) | 8
  Gene: MAGEL2 | 5
  Gene: CREBBP: number analyzed (Participants) | 1
  Gene: CREBBP | 0
  Gene: DNMT3A: number analyzed (Participants) | 1
  Gene: DNMT3A | 0
  Gene: HTR2C: number analyzed (Participants) | 3
  Gene: HTR2C | 1
  Gene: KSR2: number analyzed (Participants) | 9
  Gene: KSR2 | 3
  Gene: MRAP2: number analyzed (Participants) | 1
  Gene: MRAP2 | 0
  Gene: RPGRIP1L: number analyzed (Participants) | 3
  Gene: RPGRIP1L | 1
  Gene: TBX3: number analyzed (Participants) | 4
  Gene: TBX3 | 2
  Gene: TRPC5: number analyzed (Participants) | 2
  Gene: TRPC5 | 1

ADVERSE EVENTS:
Time Frame: Stage 1 : Baseline to Week 16 Stage 2 : Week 16 to Week 44
Description: Stage 1: Safety Analysis Set included all participants who received at least one dose of trial medication.
  Stage 2: Safety Analysis Set Enrolled in Stage 2 included all participants who were enrolled in Stage 2 and received at least one dose of trial medication in Stage 2. Three participants in the placebo group were rescued with setmelanotide open-label during Stage 2. They were classified to setmelanotide group.
Arm/Group | Stage 1: Setmelanotide (Open-Label) | Stage 2: Setmelanotide (Double-Blind) | Stage 2: Placebo (Double-Blind)
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/35 | 0/14
Serious Adverse Events (participants affected / at risk) | 6/164 | 0/35 | 0/14
Other Adverse Events (participants affected / at risk) | 160/164 | 25/35 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Setmelanotide (Open-Label) (N=164) | Stage 2: Setmelanotide (Double-Blind) (N=35) | Stage 2: Placebo (Double-Blind) (N=14)
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Setmelanotide (Open-Label) (N=164) | Stage 2: Setmelanotide (Double-Blind) (N=35) | Stage 2: Placebo (Double-Blind) (N=14)
Injection site erythema (General disorders) | 62 | 1 | 2
Injection site pain (General disorders) | 46 | 0 | 1
Injection site induration (General disorders) | 47 | 1 | 2
Injection site pruritus (General disorders) | 49 | 1 | 0
Fatigue (General disorders) | 29 | 0 | 1
Injection site oedema (General disorders) | 20 | 1 | 0
Injection site bruising (General disorders) | 22 | 0 | 0
Injection site swelling (General disorders) | 6 | 0 | 0
Injection site reaction (General disorders) | 9 | 1 | 0
Injection site discolouration (General disorders) | 10 | 0 | 0
Injection site warmth (General disorders) | 3 | 0 | 0
Pain (General disorders) | 5 | 0 | 0
Influenza like illness (General disorders) | 5 | 0 | 0
Injection site haemorrhage (General disorders) | 3 | 0 | 0
Pyrexia (General disorders) | 4 | 0 | 1
Injection site haematoma (General disorders) | 2 | 0 | 0
Peripheral swelling (General disorders) | 2 | 0 | 0
Thirst (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Crying (General disorders) | 1 | 0 | 0
Energy increased (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0
Injection site discomfort (General disorders) | 1 | 0 | 0
Injection site nodule (General disorders) | 1 | 0 | 0
Injection site urticaria (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Mucosal pigmentation (General disorders) | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0
Swelling face (General disorders) | 1 | 0 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0
Hunger (General disorders) | 0 | 1 | 1
Impaired healing (General disorders) | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 130 | 7 | 1
Ephelides (Skin and subcutaneous tissue disorders) | 7 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 10 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Nail pigmentation (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Solar lentigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Acanthosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin striae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 75 | 4 | 0
Vomiting (Gastrointestinal disorders) | 41 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 22 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 2 | 2
Pigmentation lip (Gastrointestinal disorders) | 9 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 7 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 2 | 2
Oral pigmentation (Gastrointestinal disorders) | 4 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 2 | 1 | 0
Tongue pigmentation (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gingival hyperpigmentation (Gastrointestinal disorders) | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Oral macule (Gastrointestinal disorders) | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 52 | 7 | 2
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 43 | 4 | 0
Dizziness (Nervous system disorders) | 8 | 1 | 0
Disturbance in attention (Nervous system disorders) | 2 | 0 | 0
Migraine (Nervous system disorders) | 2 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 0
Formication (Nervous system disorders) | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 14 | 4 | 1
COVID-19 (Infections and infestations) | 7 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 4 | 1 | 0
Influenza (Infections and infestations) | 5 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 2 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Libido increased (Psychiatric disorders) | 15 | 0 | 0
Disturbance in sexual arousal (Psychiatric disorders) | 11 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 0 | 0
Depression (Psychiatric disorders) | 4 | 0 | 0
Libido decreased (Psychiatric disorders) | 3 | 0 | 0
Nightmare (Psychiatric disorders) | 2 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0
Social anxiety disorder (Psychiatric disorders) | 1 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 10 | 0 | 0
Spontaneous penile erection (Reproductive system and breast disorders) | 6 | 0 | 0
Erection increased (Reproductive system and breast disorders) | 4 | 1 | 0
Clitoral engorgement (Reproductive system and breast disorders) | 2 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 0
Menstruation delayed (Reproductive system and breast disorders) | 1 | 0 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 2 | 0 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 1 | 0
Penile swelling (Reproductive system and breast disorders) | 1 | 0 | 0
Semen discolouration (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 3 | 1 | 1
Prothrombin time prolonged (Investigations) | 3 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 1
International normalised ratio increased (Investigations) | 2 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Bacterial test positive (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Cardiac stress test abnormal (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 0
High density lipoprotein decreased (Investigations) | 1 | 0 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 1 | 0 | 0
Nitrite urine present (Investigations) | 1 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 0
Red cell distribution width increased (Investigations) | 1 | 0 | 0
White blood cells urine (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1 | 1
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1
Influenza A virus test positive (Investigations) | 0 | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Urinary tract procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Mesenteric lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Urine abnormality (Renal and urinary disorders) | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 2 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Eye colour change (Eye disorders) | 1 | 0 | 0
Blepharal pigmentation (Eye disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Ocular icterus (Hepatobiliary disorders) | 1 | 0 | 0
Dental implantation (Surgical and medical procedures) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information regarding setmelanotide supplied by Rhythm to the investigator is privileged and confidential information. The investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from Rhythm. The information obtained from the clinical study will be used towards the development of setmelanotide and may be disclosed to regulatory authority(ies), other investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04963231/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT04963231/SAP_001.pdf